CLINICAL TRIAL: NCT06162715
Title: GLP-1 Receptor Agonists Post-Bariatric Surgery (GRABS) Pilot Trial
Acronym: GRABS-0
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jason Samuels, Assistant Professor of Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR72411
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-03

CONDITIONS: Severe Obesity; Obesity; BMI Greater Than 30
Keywords: bariatric surgery; Roux-en-Y Gastric Bypass; GLP-1 Receptor Agonists; Tirzepatide; Obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide Group (Experimental): Participants in the TRZ cohort will initiate a standardized dose titration as described in the package insert. Participants will begin TRZ at 2.5 mg for four weeks and then increase by 2.5 mg every 4 weeks to a maximum dose of 15 mg. If subjects experience intolerable GI symptoms, they will be allowed to decrease to a lower dose by 2.5 mg for 2 weeks, at which point another attempt at an increased dose will be trialed. Should patients not tolerate a higher dose a second time, they will have the dose again lowered by 2.5 mg and kept at the lower dose for the remainder of the study, except for patients who do not tolerate two attempts at 5 mg. For patients who fail to titrate to at least 5 mg TRZ, a third attempt at an increased dose will be attempted 4 weeks after the second decrease in dose. These patients will then remain on 5 mg for the remainder of the intervention period. All participants receiving TRZ will be pooled in terms of outcomes measures.
  Interventions: Drug: Tirzepatide
- Control - Standard of care Post-Gastric Bypass Surgery (Other): Patients randomized to the control arm will receive the standard of care for weight maintenance after gastric bypass including dietary guidance provided by the Vanderbilt Surgical Weight Loss handbook for 24 weeks. After 24 weeks, particiapnts in the control arm will crossover to the Tirzepatide arm and receive 24 weeks of TRZ following the same titration.
  Interventions: Other: Standard of Care post-gastric bypass

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide will be initiated 12 or 18 months (12 months + 24 weeks) after patients undergo Roux-en-Y Gastric Bypass. Patients will be started on the lowest dose of 2.5 mg and the dose increased every 6 weeks following an adaptive maximum dose titration protocol. Patients will then complete a final 4 weeks of the study drug.
  Other Names: Zepbound; Mounjaro
  Arms: Tirzepatide Group
Other: Standard of Care post-gastric bypass — Patients randomized to the control arm will receive the standard of care for weight maintenance after gastric bypass including dietary guidance provided by the Vanderbilt Surgical Weight Loss handbook. This includes recommendations for 64 oz of fluids per day, ≥60 grams of protein/day, and daily bariatric multivitamins. Patients will continue to have access to dedicated bariatric dietitians, advanced practice providers, and surgeons on an ad hoc basis per patients' request.
  Arms: Control - Standard of care Post-Gastric Bypass Surgery

SUMMARY:
The goal of this pilot clinical trial is to determine the effectiveness of Tirzepatide in patients with persistent obesity (BMI > 30) 12 months after bariatric surgery (Roux-en-Y Gastric Bypass). The investigators also aim to determine the frequency of side effects with Tirzepatide in this patient population. Patients who take tirzepatide 12 months after bariatric surgery will be compared to patients who continue with the current standard of care for patients who have previously undergone Gastric Bypass Surgery.

DETAILED DESCRIPTION:
Obesity affects nearly half of the U.S. population, impacting health outcomes including diabetes, cardiovascular risk, longevity, and quality of life. While bariatric surgery such as gastric bypass stands as the most effective intervention, 65% of individuals experience persistent obesity when undergoing surgical weight loss alone. Given the wide-ranging impact of obesity on health outcomes, a critical need exists to explore the efficacy of adjuvant weight loss therapies after gastric bypass surgery. Tirzepatide (TRZ), a type of glucagon-like peptide-1 receptor agonist, shows remarkable effectiveness in medical obesity with 25% weight loss after sustained therapy. However, nearly two-thirds of patients taking medications like TRZ have mild to moderate gastrointestinal (GI) symptoms, including nausea, vomiting, and abdominal pain. These medication side-effects could be a consequence of gastroparesis via vagal stimulation of the stomach, and may represent a major driver of weight loss. Limited data exist regarding use of these newer agents, such as TRZ, in patients who have undergone gastric bypass, which disrupts vagal nerves responsible for managing food transit and gastric emptying. This is a major and timely scientific gap in understanding whether gastric bypass surgery might mitigate these GI symptoms while allowing for enhanced weight loss with adjuvant TRZ use in the post-operative period. The investigators propose a pilot, phase II, open-label trial enrolling patients twelve months after gastric bypass with a nadir Body Mass Index ≥ 30 kg/m2. Study subjects will be randomized to either 24 weeks of TRZ or post-surgery standard of care. Subjects randomized to the standard of care arm will crossover to receive the intervention drug after 24 weeks of observation. Our proposal consists of two aims. First, the investigators will determine the impact of adjuvant TRZ administration on weight, total fat mass, and lean body mass in patients with a history of gastric bypass (Aim 1). Second, the investigators aim to investigate the frequency and severity of GI discomfort associated with TRZ utilizing a validated patient reported outcome questionnaire, and they will investigate the impact of TRZ on GI motility in patients with prior Gastric Bypass (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and provide informed consent.
2. BMI > 30 12 months after bariatric surgery.
3. Age > 30 and < 65
4. Patients undergoing primary Roux-en-Y Gastric Bypass

Exclusion Criteria:

1. Inability or unwillingness of a subject to give written informed consent or comply with the study protocol.
2. Diagnosis of type I Diabetes
3. Revisional bariatric surgery (prior adjustable gastric band, sleeve gastric, vertical banded gastroplasty).
4. Use of medications for type 2 di
5. Hemoglobin A1c > 8.5 in last 3 months.
6. Patient-reported Tobacco, e-cigarette, or smoked marijuana use within 12 months As this would preclude patients from undergoing bariatric surgery.
7. Personal history of pancreatitis as determined by history.
8. Personal or family history of medullary thyroid cancer by history or multiple endocrine neoplasia syndrome type 2
9. Pregnancy by urine testing, current lactation, or plans to become pregnant during the study period.
10. Use of systemic glucocorticoids in the past 28 days
11. Myocardial infarction, unstable angina, stroke, or heart failure (NYHA class II) within 1 year by history.
12. History of solid organ transplant.
13. History of physician-diagnosed malignancy (other than excised non-melanoma skin cancer) in the past 5 years.
14. Current uncontrolled hypertension (systolic >150, diastolic >90) or untreated hyperthyroidism.
15. Current, diagnosed, or self-reported drug or alcohol abuse that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements.
16. Screening creatinine elevation with EGFR < 60 at time of randomization.
17. Tobacco use in last 12 months
18. Pregnancy
19. Prisoners
20. Unable or unwilling to follow-up
21. Unable to understand English/Spanish

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss | baseline to 24 weeks
  Change in weight over time.

SECONDARY OUTCOMES:
Change in body composition | baseline to 24 weeks
  Changes in fat mass
Gastrointestinal symptoms | baseline to 24 weeks
  Gastroparesis Cardinal Symptom Index
Acetaminophen Area Under the Curve | baseline to 24 weeks
  Changes in acetaminophen area under the curve in the intervention arm
Lean body mass | 24 weeks
  Utilizing DXA, we will determine changes in lean body mass in both arms

OTHER OUTCOMES:
weight regain after TRZ discontinuation | weeks 24 to 48
  Degree of weight regain in intervention arm after discontinuation of TRZ
Obesity remission | baseline to 24 weeks
  incidence of obesity remission (BMI < 30)
Remission of pre-existing comorbidities | baseline to 24 weeks.
  Incidence of remission of Type 2 Diabetes, Hyperlipidemia, Hypertension
change in anthropometric measurements | baseline to 24 weeks
  Changes in clinical obtained anthropometric measurements including waist circumference and waist-to-hip ratio
changes in body composition | baseline to 24 weeks.
  Changes in DXA-proven body composition including lean body mass and ratio of lean body mass to fat mass
Change in PAGI-SYM sub-scale scores | baseline to 24 weeks
  1. heartburn/regurgitation, 2. nausea/vomiting, 3. postprandial fullness, 4. bloating, 5. upper and lower abdominal pain
change in PAGI-SYM scores in the TRZ arm | baseline to week 24 and week 24 to week 28 (after TRZ discontinuation)
  Determining evolution of PAGI-SYM scores across treatment in both arms and after discontinuation of TRZ in the intervetion arm.
Difference in acetaminophen AUC between groups | baseline to 24 weeks
  difference in acetaminophen AUC between Intervention and control groups
Changes in response to mixed meal tolerance test | baseline to 24 weeks
  change in intervention arm mixed meal AUC for Glucose, Insulin, and GLP-1
Medication adherence | baseline to 24 weeks
  Incidence of missed doses, patient-driven drug discontinuation, patient withdrawal in intervention arm
Adverse events and healthcare resource utilization | baseline to 48 weeks
  Incidence of adverse events including emergency department visits, hospitalizations, and reoperations

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Samuels, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All participant-level data will be preserved and shared. Shared data will be deidentified prior to sharing. Clinicaltrials.gov will document recruitment progress and final results. Study protocols will be shared with publications as supplementary data and made available upon request. All participant consent document will be collected and stored electronically utilizing the REDCap study data repository. The REDCap data warehouse will also contain the study data dictionary. Study protocols have also been published on the ClinicalTrials.gov and any protocol amendments will be reflected on the ClinicalTrials.gov study page. The investigators will utilize the Research Electronic Data Capture (REDCap) data warehouse maintained locally at Vanderbilt for all data collection. Upon study completion and prior to closing the REDCap data warehouse for this study, the investigators will archive all data after removing patient identifiers in the Open Science Framework data repository.
Supporting Information: Study Protocol, SAP
Time Frame: Per institutional policy, data will be maintained in the local REDCap data repository for 6 years after closure of the study. Following this period, data will be deidentified and uploaded to the OSF repository, which has funding for at least 50 years of data storage.

DOCUMENTS (1):
  • Informed Consent Form (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT06162715/ICF_000.pdf